CLINICAL TRIAL: NCT06466148
Title: JessieHug Feasibility and Usability Assessment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Empatica, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 23-08026420
Record Dates: First submitted 2024-06-12; First posted 2024-06-20 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: SIDS
Keywords: medical device; wearable medical device; infants
MeSH Terms: conditions — Sudden Infant Death

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- Newborn Cohort (Experimental): The JessieHug device will be placed on infants two times a week to determine usability, tolerability and safety. Clinical accuracy will be assessed in one inpatient (newborn cohort) or outpatient (2 month and 4 month cohorts) session.
  Interventions: Device: JessieHug
- 2 month Cohort (Experimental): The JessieHug device will be placed on infants two times a week to determine usability, tolerability and safety. Clinical accuracy will be assessed in one inpatient (newborn cohort) or outpatient (2 month and 4 month cohorts) session.
  Interventions: Device: JessieHug
- 4 month Cohort (Experimental): The JessieHug device will be placed on infants two times a week to determine usability, tolerability and safety. Clinical accuracy will be assessed in one inpatient (newborn cohort) or outpatient (2 month and 4 month cohorts) session.
  Interventions: Device: JessieHug

INTERVENTIONS:
Device: JessieHug — Assessment of JessieHug device when placed on infants.

SUMMARY:
The goal of this clinical trial is to evaluates the usability, tolerability, and clinical accuracy of the JessieHug device, a wearable medical device for newborns and infants that collects physiological data. The main questions it aims to answer are:

* Is the device easily usable for parents of newborns and infants?
* Is the device tolerable when worn by infants and are there any safety concerns?
* Is the device able to collect clinically accurate physiologic data compared to a FDA-cleared reference device?

Participants will:

* Place the JessieHug device on their infant two times a week and complete surveys to assess usability, tolerability and safety.
* Have one session where the JessieHug device will be worn at the same time as reference device to determine accuracy.

DETAILED DESCRIPTION:
This study evaluates the usability, tolerability, and clinical accuracy of the JessieHug device, a wearable medical device for newborns and infants that continuously collects physiological data. Three cohorts of infants will be enrolled: newborn, 2-month, and 4-month groups, with each cohort undergoing data collection over a total of eight (8) weeks. The JessieHug device will be assessed for usability and tolerability through parental surveys while the baby wears the device in home and hospital settings. Clinical accuracy of the device will be evaluated through comparison to an FDA cleared reference device in a single outpatient clinic-based data collection event.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy neonates and infants, with cohorts defined by the following age ranges:

   1. newborn (0 weeks and 0/7 days to 0 weeks and 5/7 days),
   2. 2-month (6 weeks and 0/7 days to 11 weeks and 6/7 days),
   3. 4-month (14 weeks and 0/7 days to 19 weeks and 6/7 days)
2. Born after 37 0/7 weeks of pregnancy
3. Parent or legal guardian at time of discharge is able to understand and provide consent for participation
4. Parent or legal guardian at time of discharge is willing and able to participate in study procedures for the duration of the study
5. Parent or legal guardian is fluent in English
6. Parent or legal guardian has access to the internet

Exclusion Criteria:

1. Low birth weight (< 2500g)
2. Any transfer out of the well baby nursery for increased level of care, including admission to the NICU or transitional nursery.
3. Clinical indication for prolonged postnatal hospitalization (>4 days)

Ages: 0 Months to 4 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2024-04-10 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Evaluating usability of the JessieHug measured by a System Usability Survey | Every other week for through study completion (8 weeks)
  Usability as measured by an average score of at least 68 out of 100 on the System Usability Survey (Lewis & Sauro, 2018). Lowest possible score is 0 indicating low usability and highest possible score is 100 indicating high usability. Usability surveys will include questions related to ease of use, satisfaction, and confidence when interacting with the device.
Evaluating tolerability of the JessieHug measured by the Face, Legs, Activity, Cry, and Consolability Scale (FLACC) survey, which is an observer reported outcomes (ObsRO) survey. | Every week for through study completion (8 weeks)
  Tolerability as defined as a score of 5 or less on the FLACC. Lowest possible score is 0 indicating no pain and highest possible score is 10 indicating severe pain. The FLACC scale is a behavioral pain assessment scale, validated for use in children from 2 months to 7 years of age, that is used to assess pain in children who are unable to communicate their pain verbally (Voepel-Lewis et al., 1997).
Evaluating safety of the JessieHug assessed through a survey assessing adverse events and pain. | Every week for through study completion (8 weeks)
  The qualitative safety questionnaire assesses overall tolerability of the device, satisfaction of the caregiver for the tolerability of the device, pain or adverse reactions experienced, persistence of symptoms, and the degree any potential pain or adverse reactions interfered with daily activities or sleep.
Percent caregiver completing all steps without errors | At baseline
  Ability of caregivers to follow provided instructions for unpacking and setting up the JessieHug device.

SECONDARY OUTCOMES:
Validating the clinical accuracy of the physiological parameters measured by the JessieHug (SpO2) against FDA-cleared reference devices. | One session, up to 4 hours, during study period, up to 8 weeks.
  Accuracy of the SpO2 algorithm outputs derived from JessieHug sensor data as measured by the Accuracy root-mean-square (Arms) difference between the JessieHug device measurements and the reference device measurements with passing criteria of 3.5% during no-motion conditions, respectively.
Validating the clinical accuracy of the physiological parameters measured by the JessieHug (pulse rate) against FDA-cleared reference devices. | One session, up to 4 hours, during study period, up to 8 weeks.
  Accuracy of the pulse rate algorithm outputs derived from JessieHug sensor data as measured by the Accuracy root-mean-square (Arms) difference between the JessieHug device measurements and the reference device measurements with passing criteria of 3 beats per minute (bpm)during no-motion conditions, respectively .
Validating the clinical accuracy of the physiological parameters measured by the JessieHug (respiratory rate) against FDA-cleared reference devices. | One session, up to 4 hours, during study period, up to 8 weeks.
  Accuracy of the respiratory rate algorithm outputs derived from JessieHug sensor data as measured by the Accuracy root-mean-square (Arms) difference between the JessieHug device measurements and the reference device measurements with passing criteria of 3 breaths per minute (brpm) no-motion conditions, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: James M Kim, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- NewYork Presbyterian - Weill Cornell Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No